CLINICAL TRIAL: NCT00695084
Title: Constraint-Induced Movement Therapy Trial for Progressive Multiple Sclerosis
Brief Title: Constraint-Induced (CI) Movement Therapy for Progressive Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Multiple Sclerosis Society (Other)
Responsible Party: Patricia O'Looney, National Multiple Sclerosis Society
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIMSTrial; PP1395
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment with Constraint-Induced Movement Therapy
  Interventions: Behavioral: Constraint-Induced Movement Therapy

INTERVENTIONS:
Behavioral: Constraint-Induced Movement Therapy — Intensive practice with the hemiparetic arm for 30 contact hours
  Other Names: CI Therapy

SUMMARY:
This trial will evaluate whether progressive multiple sclerosis associated with hemiparesis may benefit from Constraint-Induced Movement Therapy.

DETAILED DESCRIPTION:
Constraint-Induced Movement Therapy was developed to treat stroke hemiparesis. Due to the similarity between multiple sclerosis and stroke in terms of chronic motor deficit, this trial will attempt to determine whether multiple sclerosis may benefit similarly from Constraint-Induced Movement Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic upper extremity motor deficit due to multiple sclerosis

Exclusion Criteria:

* Relapse within 3 months of planned enrollment.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Improvement on the Motor Activity Log | One year

SECONDARY OUTCOMES:
Improvement on the Wolf Motor Function Test | Pre to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Victor W Mark, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States